CLINICAL TRIAL: NCT06422975
Title: Prospective Multicentre Observational Study of Patients Treated With Vasopressin in Critical Care Units
Brief Title: Registry of Patients in Shock Treated With Vasopressin
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Other Study IDs: VASOPRES REGISTRY
Record Dates: First submitted 2024-04-29; First posted 2024-05-21 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-04

CONDITIONS: Vasopressin Causing Adverse Effects in Therapeutic Use; Shock; Vasopressor Adverse Reaction; Vasopressin Deficiency
Keywords: Vasopressin; Shock
MeSH Terms: conditions — Shock; Diabetes Insipidus, Neurogenic; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Vasopressin — Patients treated with vasopressin

SUMMARY:
Arginine-vasopressin (AVP) is a non-catecholaminergic hormone produced in the hypothalamus and released into the circulation via the neurohypophysis. It has different actions depending on the receptors through which it acts: V1 (vasoconstriction, platelet aggregation, efferent arteriole constriction of the renal glomerulus, glycogenolysis); V2 (water reabsorption, release of von Willebrand factor and factor VIII); V3 (increased cortisol and insulin).

Septic shock is the most common cause of vasoplegic shock and its management includes control of the focus, early antibiotic therapy, volume resuscitation, vasopressor therapy, support of various organ dysfunctions, as well as monitoring and follow-up.

The Surviving Sepsis Campaign (a global initiative to improve sepsis management) recommends noradrenaline as the first line of vasopressor therapy and early addition of AVP as a second line rather than further up-titration of noradrenaline when signs of hypoperfusion persist, through its action primarily on V1.

The rationale for its use in septic shock would be:

* endogenous vasopressin deficiency present in septic shock;
* as a catecholamine-sparing strategy, reducing the side effects of catecholamines;
* its potential nephroprotective effect;
* its use should be early.

The uncertainties surrounding the use of AVP in septic shock and other types of shock are many, hence the need for this registry.

DETAILED DESCRIPTION:
The main objective is to characterise the routine clinical practice of vasopressin use in the context of shock in a multicentre observational study. By collecting clinical, analytical and echocardiographic data in a uniform manner, describing the time sequence of vasopressin and/or noradrenaline use; how long vasopressin is used; and which vasoconstrictor is more frequently withdrawn earlier: vasopressin or noradrenaline.

The secondary objectives are:

* to assess what motivated the decision to initiate AVP: type of shock, perfusion parameters, noradrenaline dose;
* to define the impact of initiating AVP on noradrenaline dose (whether the dose can be reduced or not), on cardiac function (whether echocardiographic data improve or worsen) and on perfusion data (whether laboratory and clinical data such as lactate, capillary refill time, mottling score or diuresis improve or worsen);
* estimate what is the dose range of AVP used and what is the maximum dose used in routine clinical practice;
* observe when AVP is stopped, how (abruptly or progressively);
* describe the incidence of side effects of AVP, whether it is related to the dose of AVP and the comorbidities of the patients;
* assess medium/long-term outcomes: 28- and 90-day mortality, ICU and hospital stay, days of vasopressor support, days of mechanical ventilation, days of renal replacement.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years of age who is in shock and requires the administration of vasoconstrictors, to whom vasopressin is administered in the operating theatre and/or critical care unit, according to best clinical practice.

Exclusion Criteria:

* Non-consent by patient/legal representatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in shock receiving vasopressin
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Characterise the clinical practice of vasopressin use in the context of shock in a multicentre observational study. | 90 days
  Describing the time sequence of vasopressin and/or noradrenaline use (what is initiated first) during shock

SECONDARY OUTCOMES:
Assess what prompted the decision to initiate AVP | Up to 7 days
  Assess what prompted the decision to initiate AVP: type of shock (vasoplegic, hypovolemic,...), perfusion parameters (as lactate) or noradrenaline dose (microgram/kg/minute)
Define the impact of starting AVP on noradrenaline dose | Up to 7 days
  Define the impact of starting AVP on noradrenaline dose (microgram/kg/minute)
Define the impact of starting AVP on lactate level | Up to 7 days
  Define the impact of starting AVP on lactate level (mmol/L)
Observe when AVP is discontinued and how | Up to 7 days
  Describe number of participants what AVP is discontinued first and how (abruptly or progressively)
Estimate the range of doses of AVP used | Up to 7 days
  Estimate the range of doses of AVP used and the maximum dose used in routine clinical practice.
Incidence of side effects | Up to 7 days
  Describe the incidence of side effects, whether it is related to AVP dose and patients' comorbidities.
28-day all-cause mortality | 28 days
  Death on or before study day 28
90-day all-cause mortality | 90 days
  Death on or before study day 90
Incidence of new renal replacement therapy | From onset of shock until hospital discharge, an average of 2 weeks
  New receipt of renal replacement therapy after onset of shock
Vasopressor-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of vasopressor therapy prior to day 28
Intensive care unit-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of intensive care unit admission prior to day 28.
Hospital-free days to day 28 | 28 days
  Number of days between day 28 and the end of the last period of hospital admission prior to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Raquel García Álvarez, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (24):
- Spain (24):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Cabueñes, Gijón
  - Complejo Asistencial Universitario de León, León
  - Hospital Lucus Augustus, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garcia-Alvarez R, Arboleda-Salazar R. Vasopressin in Sepsis and Other Shock States: State of the Art. J Pers Med. 2023 Oct 29;13(11):1548. doi: 10.3390/jpm13111548. PMID 38003863
- [Result] Treschan TA, Peters J. The vasopressin system: physiology and clinical strategies. Anesthesiology. 2006 Sep;105(3):599-612; quiz 639-40. doi: 10.1097/00000542-200609000-00026. PMID 16931995
- [Result] Dunser MW, Lindner KH, Wenzel V. A century of arginine vasopressin research leading to new therapeutic strategies. Anesthesiology. 2006 Sep;105(3):444-5. doi: 10.1097/00000542-200609000-00004. No abstract available. PMID 16931974
- [Result] Ramasco F, Nieves-Alonso J, Garcia-Villabona E, Vallejo C, Kattan E, Mendez R. Challenges in Septic Shock: From New Hemodynamics to Blood Purification Therapies. J Pers Med. 2024 Feb 3;14(2):176. doi: 10.3390/jpm14020176. PMID 38392609
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Result] Sharshar T, Blanchard A, Paillard M, Raphael JC, Gajdos P, Annane D. Circulating vasopressin levels in septic shock. Crit Care Med. 2003 Jun;31(6):1752-8. doi: 10.1097/01.CCM.0000063046.82359.4A. PMID 12794416
- [Result] Holmes CL, Patel BM, Russell JA, Walley KR. Physiology of vasopressin relevant to management of septic shock. Chest. 2001 Sep;120(3):989-1002. doi: 10.1378/chest.120.3.989. PMID 11555538
- [Result] Martin C, Medam S, Antonini F, Alingrin J, Haddam M, Hammad E, Meyssignac B, Vigne C, Zieleskiewicz L, Leone M. NOREPINEPHRINE: NOT TOO MUCH, TOO LONG. Shock. 2015 Oct;44(4):305-9. doi: 10.1097/SHK.0000000000000426. PMID 26125087
- [Result] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Result] Demiselle J, Fage N, Radermacher P, Asfar P. Vasopressin and its analogues in shock states: a review. Ann Intensive Care. 2020 Jan 22;10(1):9. doi: 10.1186/s13613-020-0628-2. PMID 31970567
- [Result] Gordon AC, Russell JA, Walley KR, Singer J, Ayers D, Storms MM, Holmes CL, Hebert PC, Cooper DJ, Mehta S, Granton JT, Cook DJ, Presneill JJ. The effects of vasopressin on acute kidney injury in septic shock. Intensive Care Med. 2010 Jan;36(1):83-91. doi: 10.1007/s00134-009-1687-x. Epub 2009 Oct 20. PMID 19841897
- [Result] Hamzaoui O, Goury A, Teboul JL. The Eight Unanswered and Answered Questions about the Use of Vasopressors in Septic Shock. J Clin Med. 2023 Jul 10;12(14):4589. doi: 10.3390/jcm12144589. PMID 37510705
- [Derived] Garcia Alvarez R, Ramasco F, Nieves Alonso J, Mouriz L, Rama P, Bilbao I, Perez Carbonell A, Rodenas MA, Ortega F, Vives M, Calvo CA, Taboada M, Azzam A, Merino M, Martinez F, Dominguez D, de Llano CT, Adalia R, Aguilar G, Aldecoa C, Mancha B, Reyes A, Gine M, Prendes D, Garcia Fernande C, de la Calle I, Cendrero M, Martinez Lopez A, Herrero JJ, de la Torre I, Kattan E, Hernandez G. Prospective Multicenter Observational Study of Patients in Shock Treated with Vasopressin: VASOPRES Registry Study Protocol. Rev Esp Anestesiol Reanim (Engl Ed). 2025 Aug-Sep;72(7):501768. doi: 10.1016/j.redare.2025.501768. Epub 2025 May 16. PMID 40383482